CLINICAL TRIAL: NCT05527600
Title: Development and Validation of a System Based on Digital Face Recognitation for Pain Assessment in Children's Emergency
Brief Title: Evaluation of an App Based on Artificial Intelligence for Pain Assessment in Pediatric Department
Acronym: DEF II
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21-PP-16; 2021-A02726-35 (Other: ANSM)
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: C23.888.592.612.081

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- assessment of pain in Pediatric Department: 2000 children patients admitted in emmergency department
  Interventions: Diagnostic Test: intensity of acute pain evaluation

INTERVENTIONS:
Diagnostic Test: intensity of acute pain evaluation — the facial expression of each patient will be collected from a short video of 10 seconds, follow by with the evaluation of the pain intensity.

SUMMARY:
Accurate assessment of pain in Pediatric Department is challenging. However, recent publications highlight that children do not receive optimal pain management, particularly in Emergency Departments.

An Artificial Intelligence-based tool could help physicians to optimize analgesia use.

DETAILED DESCRIPTION:
Acute pain is the reason that the majority of patients present to the Emergency Department. Multiple studies conducted over many years have demonstrated that pain is poorly managed in the Emergency Department. This phenomenon has been referred to in the Medical Literature as "Oligoanalgesia.". Morever, untreated pain can have short and long term effects in Pediatric population, including sensitisation to pain episodes in later life and can affects the Neurodevelopment of the child.

The generally accepted standard for pain assessment is self-reported; however, in preverbal children who cannot communicate their pain, age-appropriate behavioural or observational pain assessment tools are recommended. Because children are not always able to voice their feelings, they completely depend on their caregiving team for the interpretation and management of their pain and discomfort. Thus, accurately validated scales to assess pain levels are crucial. In France, the EVENDOL is the most used widely scale. The EVENDOL scale (from the French Evaluation Enfant Douleur) is used to evaluate pain in children in any situation covering a wider age group than other pain scales (birth up to seven years). Despite a large number of scales with a variety of Psychometric properties having been published in the last decades, to date, there is no criterion standard when considering the assessment of pain. As a result, children continue to be suffered pain without adequate pain management. International guidelines incorporate the need for prompt recognition of pain.

Artificial Intelligence (AI) in Medicine is booming and has already proven its worth in terms of prevention, monitoring and diagnosis. AI in this field can be used to support clinician decision making, allow curiosity-driven care, remove the need to complete mundane tasks, improve communication, and facilitate collaboration. Evaluation of the face is central to all observational pain assessment tools, as the face is highly accessible and facial expressions are considered the most encodable feature of pain Therefore.the investigators aim to develop, validate and asses a system based on Digital Face Recognitation for pain assessment in the Children's Department.

ELIGIBILITY:
Inclusion Criteria:

* Child under 18
* Informed and written consent of a parent or guardian (only 1 accompanying person allowed).

Exclusion Criteria:

* Language barrier.
* Refusal to participate by parents/children
* Sign of collapsus, or in serious clinical condition (stage I or II) requiring absolute emergency care,
* Delayed mental or staturo-ponderal development
* Facial injury or wound, presence of a bandage on the face, pre-existing facial deformity

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 2000 patients under 18 year old admitted in Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
assessment of The intensity of acute pain with the EVENDOL Scale | day 0
  The intensity of acute pain will be assessed by the current reference French methods for evaluating pain in children with the EVENDOL Scale (reference between 0 and 7 years).
assessment of The intensity of acute pain with the VAS Scale | day 0
  The intensity of acute pain will be assessed by the current reference French methods for evaluating pain in children with the VAS Scale (Age > 7 years)
the facial expression captured by short video | day 0
  a short 10-second video is collected to assess facial expression of pain in children

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Nice, Nice, CHU de NICE
  - Hopital pédiatrique Fondation Lenval, Nice

IPD SHARING:
Plan to Share IPD: No